CLINICAL TRIAL: NCT04781465
Title: Feasibility Study on an Immersive Virtual Reality Tool in the Treatment of Chronic Low Back Pain
Acronym: RIVAGE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: RIVAGE
Record Dates: First submitted 2021-03-01; First posted 2021-03-04 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Chronic Low-back Pain
Keywords: Immersive Virtual Reality

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Immersive Virtual Reality (Experimental): The patients are divided into groups of 3. Each group of patients will attend 2 days of care per week (for 4 weeks) Group N ° 1: Monday and Thursday. Group N ° 2: Tuesday and Friday.
  At each visit, the patient will participate in:
  [a "Kinesitherapy" treatment and a "Virtual Immersion" treatment] + [a "Balneotherapy treatment or an" Adapted Physical Activity treatment). Each treatment lasts 1 hour 10 minutes.
  Each patient will therefore come to the center 8 times over 1 month, or 4 hours 40 minutes a week, not counting virtual reality.
  If the groups are not full or according to the advice of the healthcare team, only one group will be selected (always 3 patients) and will attend 3 days per week.
  Interventions: Device: Immersive Virtual Reality

INTERVENTIONS:
Device: Immersive Virtual Reality — Dedicated virtual reality sessions.
  * Duration 20 minutes per session.
  * The virtual reality session will be supervised by a health professional trained in this tool after 1.5 hours of training by the team responsible for the equipment (use of the equipment, and use of the 20 minutes of VR). This supervising professional may be a doctor, an occupational therapist, a caregiver or any other health professional trained in the tool under this protocol.
  * The exercises proposed will be standardized virtual reality exercises with the same exercises for all, but adapted to the level and abilities of each patient.

SUMMARY:
Chronic low back pain is a major public health problem today, because of its prevalence and its socio-professional impact. Multiple drug or non-drug treatments exist but the pain chronicization mechanism makes the management of chronic low back pain patients difficult. Stress rehabilitation programs in specialized structures have been set up to try to improve the outcome of these patients. Likewise, home exercise is recommended. However, adherence to these exercises is generally poor. Recently, there has been a growing interest in the use of new technologies, based on the use of digital tools, in the management of pain. Thus, in patients with chronic low back pain, the attractiveness of the proposed exercise programs with new technologies, the possibility of progression in the same exercise and the possibility of customizing these exercises have been reported as being able to meet the expectations of patients. for the purpose of rehabilitation. In virtual reality, users interact in an environment simulated by a 3-dimensional computer. This technology uses multisensory resources allowing the user to feel totally immersed in the virtual environment. Virtual reality has shown a benefit in the management of pain in several indications.

In low back pain patients, pain avoidance mechanisms are put in place very early due to fear of situations or movements that may reproduce or intensify the pain. Thus, for fear of pain, individuals avoid certain movements, in particular lumbar flexion movements. This avoidance of the lumbar flexion movement actually worsens the pain phenomenon because of the musculoskeletal changes associated with it. Therefore, one of the therapeutic areas for the management of chronic low back pain would be to improve lumbar flexion capacities.

DETAILED DESCRIPTION:
Thomas JS et al evaluated the benefits of a game of virtual reality baseball on improving lumbar flexion in a randomized study (virtual reality versus control). After 3 virtual reality sessions, the 2 groups were compared, there was no difference in the improvement in lumbar flexion or in the improvement in pain, probably due to the low number of sessions offered (only 3 ). Nevertheless, the harmlessness, feasibility and safety of the game were proven here. In addition, the perception of the game was positive by the participants and there was no aggravation of pain or side effects of virtual reality.

On a larger scale and more recently, France CR and Thomas JS have shown in a randomized study of 230 patients the value of an immersive virtual reality game based on the progression of lumbar flexion compared to another game that does not improve this parameter. This was a virtual reality-based rehabilitation program, carried out over 18 weeks with 3 then 2 then 1 session (s) per week; the primary endpoint was assessment of pain and disability one week after the program. There was a sharper decrease in pain and disability with play that specifically worked lumbar flexion. The progression of lumbar flexion was correlated with the decrease in pain and disability. The authors thus showed that an immersive virtual reality game combining: a way to distract the patient's attention, a target to be reached, and a progression of the lumbar flexion exercise in the game would improve pain and pain. handicap of chronic low back pain.

Virtual reality is a distraction technique, which combines visual and auditory, allowing immersion in a virtual world through a headset that transcribes a three-dimensional image. The diversion of attention by the use of virtual reality allows the patient to immerse himself in a fictitious environment thanks to a mask on the eyes that inhibits the vision of the outside world and a hearing headset reducing external sounds and reinforcing the mechanism of 'immersion. Our hypothesis is that the use of an immersive virtual reality tool would improve the rehabilitation care and the future of chronic low back pain patients, via this immersion capacity.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman whose age ≥ 18 years and <60 years
* French-speaking patient
* Affiliated with social security or, failing that, with another health insurance system.
* Non-specific low back pain +/- radiculalgia, mechanical, evolving for at least 3 months
* Patient able to understand and respond to simple instructions
* Numerical assessment scale for lumbar pain greater than or equal to 4/10
* Patient having given free, informed and express consent.

Exclusion Criteria:

* Pregnant or breastfeeding woman
* Patients with nausea, vomiting, dizziness
* Visual disturbance or hearing impairment, vestibular disorder or other disorder which, according to the investigator, makes it impossible to use a virtual reality mask or headset
* Concomitant monitoring of another rehabilitation process (physiotherapy, occupational therapy, osteopathy, or other)
* Patients with a history of neurological disorders such as epilepsy
* Major cervical or lumbar osteoarthritis or severe scoliosis making it impossible to mobilize the spinal segment concerned
* Biological inflammatory syndrome or inflammatory nature of pain
* Fibromyalgia / chronic diffuse pain syndrome
* Psychiatric pathology, except depression if the disease is controlled
* Symptomatic back pain due to neoplasia / infection / underlying vertebral fracture
* Recent spine surgery <6 months
* Active neoplasia
* Refusal to follow the entire rehabilitation program
* Geographical distance not allowing travel to a rehabilitation center
* Spinal infiltration less than 1 month old
* Patient under guardianship or curatorship
* Patient deprived of liberty
* Patient under legal protection.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2020-01-07 (Actual); Primary Completion 2021-09-06 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
To assess attendance of a rehabilitation program for chronic low back pain patients integrating immersive virtual reality sessions | Week 4
  Patient attendance to an immersive virtual reality program
To assess adherence of a rehabilitation program for chronic low back pain patients integrating immersive virtual reality sessions | Week 4
  Patient adherence to an immersive virtual reality program

SECONDARY OUTCOMES:
To evaluate patient satisfaction with the progress of the program | Week 4
  Satisfaction assessed by questionnaire
To evaluate stakeholder satisfaction with the progress of the program | Week 4
  Satisfaction assessed by questionnaire
Evaluate the improvement in pain | Day 1
  Numerical pain rating scale (0 : no pain / 10 : very strong pain)
Evaluate the improvement in pain | Week 4
  Numerical pain rating scale (0 : no pain / 10 : very strong pain)
Evaluate the overall improvement of the patient | Day 1
  Overall assessment scale for the pathology by the patient (0 : very unhappy -10 : very satisfied)
Evaluate the overall improvement of the patient | Week 4
  Overall assessment scale for the pathology by the patient (0 : very unhappy -10 : very satisfied)

CONTACTS AND LOCATIONS:
Overall Officials: Agnès PORTIER, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint-Joseph, Paris, Île-de-France Region, France